CLINICAL TRIAL: NCT05632614
Title: The Efficacy of Inspiratory Muscle Strength Training on Coronary Blood Flow in Patients With Coronary Artery Disease
Brief Title: Blood Flow Reserve: Effects After Training With Heavy Inspiratory Exercises
Acronym: BREATHE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20220463-01H
Record Dates: First submitted 2022-10-12; First posted 2022-11-30 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Disease
Keywords: inspiratory muscle strength training; coronary artery disease; positron emission tomography; myocardial blood flow
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity IMST (Active Comparator): Participants who will be trained with high-intensity IMST
  Interventions: Device: High-intensity IMST
- Low-intensity IMST (Sham Comparator): Participants who will be trained with low-intensity IMST
  Interventions: Device: Low-intensity IMST

INTERVENTIONS:
Device: High-intensity IMST — Participants will use the POWERbreathe KHP2 inspiratory muscle training device. All participants will be assigned to perform 30 inspiratory maneuvers (5 sets of 6, 1-minute rest between sets), 6 days per week, for 6 weeks. Participants will be trained at 55% PIMAX during week 1, 65% PIMAX during week 2, and 75% PIMAX during weeks 3 to 6.
  Arms: High-intensity IMST
Device: Low-intensity IMST — Participants will use the POWERbreathe KHP2 inspiratory muscle training device. All participants will be assigned to perform 30 inspiratory maneuvers (5 sets of 6, 1-minute rest between sets), 6 days per week, for 6 weeks. Participants will be trained at 15% PIMAX for 6 weeks.
  Arms: Low-intensity IMST

SUMMARY:
The goal of this single-site, parallel-group, double-blind, sham-controlled randomized control trial is to examine the effect of high-intensity inspiratory muscle strength training (IMST) on coronary blood flow assessed using positron emission tomography coronary perfusion imaging in patients with coronary artery disease (CAD).

The main question it aims to answer are:

• if high-intensity IMST will improve coronary blood flow in patients with CAD, which could be assessed using positron emission tomography coronary perfusion imaging.

Participants will be asked to complete the 8-week high-intensity or low-intensity IMST. Researchers will compare high and low-intensity IMST groups to see if coronary blood flow increases after IMST.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is a leading cause of morbidity and mortality. With the aging population, increasing number of patients with CAD has frailty and immobility. The health benefits of traditional aerobic exercise have been well-established; however, alternative exercise programs, such as inspiratory muscle training (IMST), may provide greater merits. IMST is a form of exercise that engages the diaphragm and accessory respiratory muscles to repeatedly inhale against resistance, which can be achieved in less time and widely applicable even for immobile or frail patients compared to conventional aerobic exercise. Since barriers to conventional exercise training include immobility, lack of time, and access to facilities, IMST may be a beneficial exercise form that can overcome those factors. A previous study has shown that high-intensity IMT can lower blood pressure and improved vascular endothelial function. Improvements in endothelial function of coronary arteries could improve coronary blood flow, leading to the improvement of anginal symptoms as well as quality of life. IMST might offer a widely applicable, feasible, time-efficient form of training for CAD patients. Our study will examine the preliminary efficacy of IMST on coronary blood flow in patients with CAD.

ELIGIBILITY:
Inclusion criteria:

1. ≥18 years of age;
2. Patients referred to PET at the University of Ottawa Heart Institute;
3. able to perform a respiratory exercise testing; and,
4. Patients with clinical stability, including no change in medications for the past one month.

Exclusion criteria:

1. unstable angina or established diagnosis of severe valvular heart disease, hypertrophic obstructive cardiomyopathy, chronic obstructive pulmonary disease;
2. unable to follow training/breathing instructions;
3. unable to return for follow-up visit;
4. presence of any major non-cardiac problem that would adversely affect survival during the study in the opinion of the investigator; or,
5. unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Global myocardial flow reserve | Through study completion, an average of 8 weeks
  Change in global myocardial flow reserve on positron emission tomography coronary perfusion imaging before and after IMST
Global stress myocardial blood flow | Through study completion, an average of 8 weeks
  Change in global stress myocardial blood flow on positron emission tomography coronary perfusion imaging before and after IMST

SECONDARY OUTCOMES:
Global rest myocardial blood flow | Through study completion, an average of 8 weeks
  Change in global rest myocardial blood flow on positron emission tomography coronary perfusion imaging before and after IMST
Maximum myocardial flow reserve | Through study completion, an average of 8 weeks
  Change in maximum myocardial flow reserve on positron emission tomography coronary perfusion imaging before and after IMST
Maximum myocardial blood flow at rest and stress | Through study completion, an average of 8 weeks
  Change in maximum myocardial blood flow at rest and stress on positron emission tomography coronary perfusion imaging before and after IMST
Global coronary vascular resistance at stress and rest | Through study completion, an average of 8 weeks
  Change in global coronary vascular resistance at stress and rest on positron emission tomography coronary perfusion imaging before and after IMST
Maximum coronary vascular resistance at stress and rest | Through study completion, an average of 8 weeks
  Change in maximum coronary vascular resistance at stress and rest on positron emission tomography coronary perfusion imaging before and after IMST
Mean segmental (17-segment model) myocardial flow reserve | Through study completion, an average of 8 weeks
  Change in mean segmental (17-segment model) myocardial flow reserve on positron emission tomography coronary perfusion imaging before and after IMST
Mean segmental (17-segment model) myocardial blood flow at stress and rest | Through study completion, an average of 8 weeks
  Change in mean segmental (17-segment model) myocardial blood flow at stress and rest on positron emission tomography coronary perfusion imaging before and after IMST
Maximal segmental (17-segment model) myocardial blood flow at stress and rest | Through study completion, an average of 8 weeks
  Change in maximal segmental (17-segment model) myocardial blood flow at stress and rest on positron emission tomography coronary perfusion imaging before and after IMST
Summed stress score, summed rest score, and summed difference score | Through study completion, an average of 8 weeks
  Change in summed stress score, summed rest score, and summed difference score on positron emission tomography coronary perfusion imaging before and after IMST
% left ventricular ischemia | Through study completion, an average of 8 weeks
  Change in % left ventricular ischemia on positron emission tomography coronary perfusion imaging before and after IMST
General quality of life | Through study completion, an average of 8 weeks
  Change in general Quality of life assessed using the EQ5D-5L
Angina symptom | Through study completion, an average of 8 weeks
  Change in angina symptom assessed using the Seattle angina Questionnaire
Adherence of IMST program | Through study completion, an average of 8 weeks
  The proportion of participants adhering to prescribed IMST sessions
Respiratory Muscle Strength | Through study completion, an average of 8 weeks
  Respiratory Muscle Strength assessed by % change in maximal inspiratory pressure
Resting blood pressure | Through study completion, an average of 8 weeks
  Resting blood pressure measured in a seated position after a 5-minute rest period using an automated blood pressure monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Chow, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization. Global health estimates 2020: Global cause of death, 2000-2016. World Health Organization, Geneva December 2020.
- [Background] Lee IM, Shiroma EJ, Lobelo F, Puska P, Blair SN, Katzmarzyk PT; Lancet Physical Activity Series Working Group. Effect of physical inactivity on major non-communicable diseases worldwide: an analysis of burden of disease and life expectancy. Lancet. 2012 Jul 21;380(9838):219-29. doi: 10.1016/S0140-6736(12)61031-9. PMID 22818936
- [Background] Arnett DK, Blumenthal RS, Albert MA, Buroker AB, Goldberger ZD, Hahn EJ, Himmelfarb CD, Khera A, Lloyd-Jones D, McEvoy JW, Michos ED, Miedema MD, Munoz D, Smith SC Jr, Virani SS, Williams KA Sr, Yeboah J, Ziaeian B. 2019 ACC/AHA Guideline on the Primary Prevention of Cardiovascular Disease: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2019 Sep 10;74(10):1376-1414. doi: 10.1016/j.jacc.2019.03.009. Epub 2019 Mar 17. PMID 30894319
- [Background] Warburton DE, Katzmarzyk PT, Rhodes RE, Shephard RJ. Evidence-informed physical activity guidelines for Canadian adults. Can J Public Health. 2007;98 Suppl 2:S16-68. PMID 18213940
- [Background] Kelly S, Martin S, Kuhn I, Cowan A, Brayne C, Lafortune L. Barriers and Facilitators to the Uptake and Maintenance of Healthy Behaviours by People at Mid-Life: A Rapid Systematic Review. PLoS One. 2016 Jan 27;11(1):e0145074. doi: 10.1371/journal.pone.0145074. eCollection 2016. PMID 26815199
- [Background] Chiappa GR, Roseguini BT, Vieira PJ, Alves CN, Tavares A, Winkelmann ER, Ferlin EL, Stein R, Ribeiro JP. Inspiratory muscle training improves blood flow to resting and exercising limbs in patients with chronic heart failure. J Am Coll Cardiol. 2008 Apr 29;51(17):1663-71. doi: 10.1016/j.jacc.2007.12.045. PMID 18436118
- [Background] Cipriano GF, Cipriano G Jr, Santos FV, Guntzel Chiappa AM, Pires L, Cahalin LP, Chiappa GR. Current insights of inspiratory muscle training on the cardiovascular system: a systematic review with meta-analysis. Integr Blood Press Control. 2019 May 20;12:1-11. doi: 10.2147/IBPC.S159386. eCollection 2019. PMID 31190975
- [Background] Craighead DH, Heinbockel TC, Freeberg KA, Rossman MJ, Jackman RA, Jankowski LR, Hamilton MN, Ziemba BP, Reisz JA, D'Alessandro A, Brewster LM, DeSouza CA, You Z, Chonchol M, Bailey EF, Seals DR. Time-Efficient Inspiratory Muscle Strength Training Lowers Blood Pressure and Improves Endothelial Function, NO Bioavailability, and Oxidative Stress in Midlife/Older Adults With Above-Normal Blood Pressure. J Am Heart Assoc. 2021 Jul 6;10(13):e020980. doi: 10.1161/JAHA.121.020980. Epub 2021 Jun 29. PMID 34184544
- [Background] Craighead DH, Heinbockel TC, Hamilton MN, Bailey EF, MacDonald MJ, Gibala MJ, Seals DR. Time-efficient physical training for enhancing cardiovascular function in midlife and older adults: promise and current research gaps. J Appl Physiol (1985). 2019 Nov 1;127(5):1427-1440. doi: 10.1152/japplphysiol.00381.2019. Epub 2019 Sep 26. PMID 31556835
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564